CLINICAL TRIAL: NCT03923972
Title: Exercise Training and Physical Rehabilitation in Patients With Chronic Kidney Disease in Europe - What is the Problem? - A European Survey Study
Brief Title: Exercise Training and Physical Rehabilitation in Patients With Chronic Kidney Disease in Europe - What is the Problem?
Acronym: EUSUREX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Skane University Hospital (Other)
Collaborators: Cardenal Herrera University (Other); Aristotle University Of Thessaloniki (Other); Queen Margaret University (Other); Universiteit Antwerpen (Other); Tartu University Hospital (Other); University of Pisa (Other); King's College London (Other); Sozialstiftung Bamberg (Other); Azienda Ospedaliera Bianchi-Melacrino-Morelli (Other)
Responsible Party: Principal Investigator, Naomi Clyne, associate professor, Skane University Hospital
Other Study IDs: EUSUREX-01
Record Dates: First submitted 2019-03-12; First posted 2019-04-23 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Renal Insufficiency, Chronic; Kidney Failure, Chronic; Exercise
Keywords: physical activity; exercise training; surveys and questionnaires; chronic kidney disease; dialysis; kidney transplantation; health care facilities
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with chronic kidney disease: Patients with non dialysis dependent chronic kidney disease stages 4-5, patients on renal replacement therapy treated with peritoneal dialysis or hemodialysis, patients after renal transplantation
- Nephrologists: physicians treating patients with chronic kidney disease
- Nephrology nurses: nurses caring for patients with chronic kidney disease
- heads of Nephrology departments: Medical and/or administrative directors of e nephrology department with knowledge of the healthcare system in their country

SUMMARY:
This study evaluates possible barriers to physical activity/exercise training for patients with chronic kidney disease in Europe. The study's aim is to investigate structural problems and attitudes at different levels of care. Both a systemic and individual approach are applied. Barriers due to health care organisation and reimbursement policies will be investigated in the health care system and at the renal unit. Perceived benefits of physical activity and personal attitudes towards a healthy lifestyle will be investigated in nephrologists and renal nurses. Patients' health related quality of life, attitudes and perceived availability will be explored.

DETAILED DESCRIPTION:
Exercise training and physical rehabilitation in patients with chronic kidney disease in Europe - what is the problem? - A European survey study -EUSUREX (EUropean SUrvey on Renal EXercise)

Purpose Firstly, to identify potential barriers for integrating exercise training into regular therapy for patients with chronic kidney disease in different European countries.

Secondly, to use this knowledge of the importance of different barriers to promote the use of exercise training as therapy and to target the respective levels.

Thirdly, if there are obvious differences at the level of the health care system, positive examples from one country could be used as a lever in another country.

Background Lack of physical activity is common in patients with chronic kidney disease (CKD) and is a risk factor for increased mortality (1) as in the general population (2). To date there is a body of scientific evidence showing that patients with nondialysis dependent CKD, patients on maintenance dialysis and patients after renal transplantation all benefit from regular exercise training (3,4).

Many national societies worldwide recommend that exercise training be incorporated into treatment of patients with CKD. A number of qualitative and quantitative studies have highlighted various barriers to exercise training (5-12). The most commonly described barriers include patient hesitation due to feeling tired, not having time, being in pain or just being afraid to move. Other common barriers are staff related. Nurses are pressed for time and do not feel they have knowledge or competence to assist patients. Nephrologists do not ask patients about their physical activity or just do not think it is important. Some studies, albeit in general practitioners and cardiologists, have shown an association between the physicians' own level of physical activity and propensity to recommend physical activity to their patients. In a pilot study, the investigators found association between both renal physicians and nurses levels of physical activity and propensity to recommend physical training to their patients with chronic kidney disease (13).

No study has to date described possible barriers due to the health care system. These could be caused by the remuneration system, traditions pertaining to employing dedicated and specially trained physiotherapists or exercise physiologists or other causes.

There is to the investigators' knowledge no study employing a European perspective and investigating patients', physicians', nursing staff's and hospital administrators' attitudes and perception of barriers to integrating regular exercise training into routine clinical care. Nor is there any study examining the whole spectrum of chronic kidney disease, i.e comprising nondialysis dependent CKD, maintenance dialysis treatment, including both patients treated with hemodialysis and peritoneal dialysis, and after renal transplantation.

Methods Selection of participating centres with research subjects and patients A list of all Renal units for each country was sent to professor Carmine Zoccali's group with headquarters in Reggio di Calabria, where dr Giovanni Tripepi, head biostatistician of the CNR-IFC Clinical Epidemiology and Pathophysiology of Renal Diseases and Hypertension Unit, randomly selected one renal unit per 4 million inhabitants.

The investigators aim is to include at least 1000 patients. If the investigators do not receive a sufficient number of replies from the patients from the centres the investigators have already contacted (all randomly selected), the investigators will make another random selection in the various countries and involve (just for the Patient questionnaire) other centres.

Construction of the questionnaires Step 1. National experts interested in the field of exercise training in patients with CKD were consulted.

Step 2. Current literature, pre-existing questionnaires and general experiences and suggestions received by various colleagues were collected and formed a basis for constructing the questionnaires.

Step 3. Five questionnaires were constructed targeting country level organization of physical rehabilitation programs as well as clinicians', nurses' and patients' perception about physical exercise and physical rehabilitation programmes.

1. Country level questionnaire - general questions about physical rehabilitation opportunities at country level,
2. Renal unit level questionnaire - questions about physical rehabilitation programs at the renal unit level,
3. Nephrologist questionnaire - questions about how the problem is perceived by clinicians
4. Nurse questionnaire - questions about how the problem is perceived by nurses
5. Patient questionnaire - the SF-36 was used with added questions about how the problem is perceived by the patients.

Step 4 Questionnaires were validated for clarity and consistency of content in randomly selected units in EU countries.

Validation questions were constructed for each questionnaire. Each participating country has one or two national leaders responsible for the study.

The national leaders sent the questionnaires 2, 3 and 4 together with corresponding validation questionnaires to the heads of the randomly selected Renal units in their respective countries for validation by the head of the unit, the physicians and head nurse(s). Questionnaires 1 and 5 were validated by each country's national leader.

Step 5 After validation the questionnaires were once again sent to the national leaders for distribution to each country's randomly selected renal centres for a new evaluation to ensure that the questionnaires are clear and are consistent with content. Further refinements if necessary will be performed after which the final step of validation is completed. Finally, each national leader will translate the appropriate questionnaires as deemed necessary. The SF-36 is translated and validated in most European languages. The national leader will only need to translate the additional questions.

Distribution of questionnaires Once the questionnaires have been validated and unanimously approved, the colleagues at the various centres involved in the validation process (all randomly selected) will be asked to compile the VALIDATED Country-, Renal Unit-, Clinician-, Nurse- questionnaires and administer the Patient questionnaire to the whole (consenting) patient population at their respective centres.

Statistical evaluation The questionnaires will be sent to CNR-IFC Clinical Epidemiology and Pathophysiology of Renal Diseases and Hypertension Unit in Reggio di Calabria for statistical evaluation. Data description and data analysis will be performed with parametric and non-parametric methods recommended for the analysis of questionnaires (14) by the STATA 15 statistical package.

ELIGIBILITY:
Inclusion Criteria:

* all adult patients with non-dialysis dependent chronic kidney disease, peritoneal dialysis, hemodialysis, renal transplantation
* all active physicians in the department of nephrology involved in patient care
* all active nurses in the department of nephrology involved in patient care
* all heads of nephrology departments

Exclusion Criteria:

* children
* no physical disability making it impossible to conduct exercise training
* no mental disability or language problem making it impossible to understand and fill in a questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease comprising non dialysis dependent patients with stages 4-5, patients on peritoneal or hemodialysis, after a renal transplantation, physicians and nurses involved in the treatment of these patients and the director responsible for managing the nephrology department.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Exercise prescription to patients with chronic kidney disease | through study completion, an average of one year
  Number of units with exercise prescription plans
Nephrologists exercise habits | through study completion, an average of one year
  Number of nephrologists participating in regular exercise
Renal nurses exercise habits | through study completion, an average of one year
  Number of renal nurses participating in regular exercise
CKD patients exercise habits | through study completion, an average of one year
  Number of patients who have received prescription of exercise training
Health related quality of life in patients with CKD | through study completion, an average of one year
  SF-36 quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Carmine Zoccali, MD, PhD, Study Chair — CNR-IFC Clinical epidemiology of renal diseases and hypertension, Reggio Cal.; Naomi Clyne, MD, PhD, Study Chair — Clinical Sciences, Lund, Lund University and Skåne University Hospital; Carmine Zoccali, MD, PhD, Principal Investigator — CNR-IFC Clinical epidemiology of renal diseases and hypertension; Francesca Malamacci, MD, PhD, Principal Investigator — Azienda Ospedaliera Bianchi-Melacrino-Morelli di Reggio Calabria; Naomi Clyne, MD, PhD, Principal Investigator — Clinical Sciences, Lund, Lund University and Skåne University Hospital; Evangelia Kouidi, MD, PhD, Principal Investigator — Aristotle University Of Thessaloniki; Amaryllis VanCraenenbroeck, MD, PhD, Principal Investigator — KU Leuven; Adamasco Cupisti, MD, PhD, Principal Investigator — University of Pisa; Clemens Grupp, MD, PhD, Principal Investigator — Sozialstiftung Bamberg; Mai Rosenberg, MD, PhD, Principal Investigator — University of Tarttu
Locations (2):
- Sweden (2):
  - Hallands sjukhus, Halmstad
  - Ljungby lasarett, Ljungby

IPD SHARING:
Plan to Share IPD: No